CLINICAL TRIAL: NCT05367960
Title: An Open-Label Extension Study of BPN14770 in Subjects With Fragile X Syndrome
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Tetra Discovery Partners (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPN14770-CNS-302
Record Dates: First submitted 2022-04-29; First posted 2022-05-10 (Actual); Last update posted 2025-10-03 (Actual); Status verified 2025-10

CONDITIONS: Fragile X Syndrome
MeSH Terms: conditions — Fragile X Syndrome | interventions — BPN14770

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Study Drug (BPN14770) (Other): 25mg BID Study Drug BPN14770 (Adults) or 15mg BID Study Drug BPN14770 (Adolescents with body weight <43 kg)
  Interventions: Drug: Zatolmilast/ BPN14770

INTERVENTIONS:
Drug: Zatolmilast/ BPN14770 — 25mg zatolmilast/BPN14770 (Adults) or 15 mg zatolmilast/BPN14770 (Adolescents <43 kg)

SUMMARY:
This is a 4-year, open-label extension (OLE) study for subjects completing one of two double-blind clinical trials with BPN14770, Study BPN14770-CNS-301 (in adult males) and Study BPN14770-CNS-204 (in adolescent males).

DETAILED DESCRIPTION:
This is a 4-year open-label extension (OLE) study for subjects completing one of two double-blind clinical trials with BPN14770, Study BPN14770-CNS-301 (in adult males) and Study BPN14770-CNS-204 (in adolescent males). The primary objective of this OLE is to assess the long-term safety and tolerability of BPN14770 in these subjects with fragile X syndrome (FXS) who were treated in one of those parent clinical trials.

ELIGIBILITY:
Inclusion Criteria:

1. Subject has completed the Week 13 visit, whether on treatment or discontinued from treatment, from one of two parent clinical trials with

   BPN14770:
   1. Study 204
   2. Study 301 Subjects who discontinued study treatment early due to AEs deemed related to study treatment by the investigator in one of the parent studies will NOT be eligible, regardless of whether the Week 13 visit was completed.
2. Subjects with a history of seizure disorder who are currently receiving treatment with antiepileptics must have remained seizure-free during the parent study. Any subject experiencing a seizure during the parent study is not eligible to continue into this long-term safety study.
3. Subject must be willing to practice barrier methods of contraception while on study, if sexually active. Abstinence is also considered a reasonable form of birth control in this study population.
4. Subject has a parent, legal authorized guardian, or consistent caregiver.
5. Subject and caregiver are able to attend the clinic regularly and reliably.
6. If subject is his own legal guardian, he is able to understand and sign an informed consent form to participate in the study.
7. For subjects who are not their own legal guardian, subject's parent/legally authorized guardian is able to understand and sign an informed consent form for their child to participate in the study.
8. If subject is not his own legal guardian, subject must provide assent for participation in the study if he has the cognitive ability to do so.

Exclusion Criteria:

* 1. History of, or current cardiovascular, renal, hepatic, respiratory, gastrointestinal, psychiatric, neurologic, cerebrovascular, or other systemic disease that would place the subject at risk or potentially interfere with the interpretation of the safety, tolerability, or efficacy of the study treatment. Common conditions such as mild hypertension, etc. are allowed per the principal investigator's (PI) judgement as long as they are stable and controlled by medical therapy that is constant for at least 4 weeks before randomization.

  2. Renal impairment, defined as serum creatinine >1.25×ULN per the latest available laboratory results from the parent study.

  3. Cirrhosis, unstable chronic liver disease or acute liver disease. Hepatic impairment, defined as ALT or AST elevation > 2 × ULN per the latest available laboratory results from the parent study. Subjects with stable chronic hepatitis B on oral anti-viral therapy and subjects cured of chronic hepatitis C are allowed. Subjects with Gilbert syndrome are allowed.

  4. Clinically significant abnormalities, in the investigator's judgement, in safety laboratory tests, vital signs, or ECG, as measured at the final visit of the parent study.

  5. Substance abuse documented during the parent study.

  6. Significant hearing or visual impairment that may affect the subject's ability to complete the test procedures.

  7. Concurrent major psychiatric condition (eg, major depressive disorder, schizophrenia, or bipolar disorder) as confirmed by the investigator. Subjects with additional diagnosis of autism spectrum disorder or anxiety disorder will be allowed.

  8. Subject has active diseases that would interfere with participation, such as acquired immunodeficiency disorder, hepatitis C, hepatitis B, or tuberculosis.

  9. Subject has participated in another clinical trial within the 30 days preceding screening OTHER THAN one of the two studies required per Inclusion Criteria 1.

Ages: 9 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — Male
Enrollment: 314 (Actual)
Dates: Start 2022-11-01 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability of BPN14770 | 24 months
  Long-term safety and tolerability of BPN14770 in these subjects with fragile X syndrome (FXS) who were treated in one of those parent clinical trials. Safety/tolerability endpoint: Treatment Emergent Adverse Events (TEAEs), which will be coded using the Medical Dictionary for Regulatory Activities. Subject incidence of each system organ class and unique preferred term will be tabulated, including all TEAEs, at least possibly related TEAEs, TEAEs resulting discontinuation of study treatment, TEAEs by intensity, and treatment-emergent SAEs. The safety analysis will be descriptive in nature.

SECONDARY OUTCOMES:
National Institute of Health (NIH)- Toolbox Cognitive Battery (TCB) | 24 Months
  National Institute of Health (NIH)- Toolbox Cognitive Battery (TCB):
  cognitive battery assessing cognition from baseline to week 6, 12, 24, 26, 52 in the NIH-TCB CCC, which is calculated from the Picture Vocabulary and Oral Reading domains.
Numerical rating scale scores (NRS) scores | 24 Months
  Numerical rating scale scores (NRS) scores: parent(s), legal authorized guardian(s), or consistent caregiver(s)-rated assessment of subject-specific behavioral anchors for domains of Daily Function, Language, Academic Skills (subjects from Study 204 only), and Emotions/Behaviors versus Baseline The 3 subject-specific behaviors per domain, as selected by the caregiver in the parent study, will be used for rating throughout the clinical trial. For each of the 3 behaviors chosen within each domain, the parent(s), legal authorized guardian(s), or consistent caregiver(s) will rate the individual from 0 "worst problem" to 10 "no problem at all" so that improvements or worsening in the specific behavior over the treatment period can be evaluated. The caregiver completing the assessment should remain the same at all applicable visits throughout the trial.
Caregiver Global Impression of Improvement (CaGI-I) assessments: | 24 Months
  Caregiver Global Impression of Improvement (CaGI-I) assessments: for the general domains of Daily Function, Language, Academic Skills (subjects from Study 204 only), and Emotions/Behaviors versus baseline. The CaGI-I is a global measure to provide a caregiver's perspective of a subject's overall condition. The assessment of improvement is a 7-point scale that requires the caregiver to assess how much the subject's illness has improved or worsened relative to a baseline state (Week 13 of the parent study) at the beginning of the intervention, and rated as: 1, very much better; 2, much better; 3, a little better; 4, no change; 5, a little worse; 6, much worse; or 7, very much worse.
Clinical Global Impression Severity (CGI-S) assessments: | 24 Months
  Clinical Global Impression Severity (CGI-S) assessments: for general domains of Daily Function, Language, Academic Skills (subjects from Study 204 only), and Emotions/Behaviors versus baseline. In this study, the general domains of Daily Function, Language, Academic Skills (Study 204 subjects only), and Emotions/Behaviors will be assessed using the CGI-S and CGI-I assessment tools. The assessment of severity will be made with a 7-point scale: 1, none; 2, very mild; 3, mild; 4, moderate; 5, marked; 6, severe; 7, extremely severe. The comparison will be made with respect to the overall experience of the clinician with individuals of the same age and sex. In this study, the general domains of Daily Function, Language, Academic Skills (Study 204 subjects only), and Emotions/Behaviors will be assessed. The CGI-S must be administered by the same rater for a given subject at all applicable visits throughout the trial.
Vineland-3 Adaptive Behavior Scale (Vineland-3) | 24 Months
  Vineland-3 Adaptive Behavior Scale (Vineland-3): clinician-administered comprehensive interview yielding adaptive behavior composite score and domain standard scores in domains of communication (receptive, expressive, and written adaptive language functions), daily living skills (personal, domestic, and community skills), and socialization (interpersonal relationships, play and leisure time, and coping abilities) versus baseline. The Vineland-3 is a clinician-administered comprehensive interview yielding adaptive behavior composite score and domain standard scores in domains of: Communication (receptive, expressive, and written adaptive language functions); Daily Living Skills (personal, domestic, and community skills); and Socialization (interpersonal relationships, play and leisure time, and coping abilities) (Pepperdine 2017).
Verbal Knowledge Test from the Stanford-Binet (ed 5) IQ assessment | 24 Months
  Verbal Knowledge Test from the Stanford-Binet (ed 5) IQ assessment versus baseline.
  The Verbal Knowledge test is a specific subtest within the SB-5 instrument. This test asks an individual to define everyday words. A full SB-5 assessment of IQ obtained anytime in the 6 months before Day 1 may have been used, provided that individual items scores or z-deviation scores for each item were available. If the required assessment was not available in this time frame, the full SB-5 assessment was completed within the screening window and prior to conducting the NIH-TCB assessments at screening. The same screening SB-5 used in the parent study should be used for the screening assessment in this OLE study. The SB-5 subtest for Verbal Knowledge test does not need be performed at screening, since the results from the parent study is available; the Verbal Knowledge test must be performed at Week 52/early termination.
Aberrant Behavior Checklist (ABC) scores | 24 Months
  Aberrant Behavior Checklist (ABC) scores: parent(s), legal authorized guardian(s), or consistent caregiver(s)-rated scale with six subscales to assess irritability, lethargy, hyperactivity, inappropriate speech, and social avoidance, using the FXS-specific factoring system (ABC-FX) versus baseline. The ABC is a 58-item parent(s), legal authorized guardian(s), or consistent caregiver(s) rating scale used to assess behaviors in FXS across 6 dimensions or subscales: inappropriate speech, irritability, hyperactivity, lethargy/withdrawal, stereotypy, and social avoidance (Sansone 2012).
  Items are evaluated on a 4-point Likert scale ranging from 0 (not at all a problem) to 3 (the problem is severe in degree). This scale has been used extensively in FXS in clinical trials and other projects. The ABC will be scored using the FXS-specific factoring system (ABC-FX). The caregiver completing the assessment should remain the same at all applicable visits throughout the trial.
Anxiety, Depression, and Mood Scale (ADAMS) scores | 24 Months
  Anxiety, Depression, and Mood Scale (ADAMS) scores: parent(s), legal authorized guardian(s), or consistent caregiver(s)-rated scale with a total score and six subscores to assess inappropriate speech, irritability, hyperactivity, lethargy/withdrawal, stereotypy, and social avoidance versus baseline. The ADAMS is a 28-item behavior-based informant instrument rated by the parent(s), legal authorized guardian(s), or consistent caregiver(s). The scale is composed of 5 factors, which address Manic/Hyperactive Behavior, Depressed Mood, Social Avoidance, General Anxiety, and Obsessive/Compulsive Behavior. A caregiver identified upon enrollment of subject should have intimate knowledge of the subject's situation and level of impairment to be able to provide accurate information as required to complete the ADAMS. The caregiver completing the assessment should remain the same at all applicable visits throughout the trial.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Berry-Kravis, MD, Principal Investigator — Rush University Medical Center
Locations (17):
- United States (17):
  - Amnova Clinical Research, Irvine, California
  - Thompson Autism & Neurodevelopment Center - CHOC, Orange, California
  - MIND Institute UC Davis Medical Center, Sacramento, California
  - Children's Hospital Colorado, Aurora, Colorado
  - University of Miami, Miami, Florida
  - Emory University School of Medicine, Atlanta, Georgia
  - Rush University Medical Center, Chicago, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Boston Children's Hospital, Boston, Massachusetts
  - U Mass, Worcester, Massachusetts
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Suburban Research Associates, Media, Pennsylvania
  - Clinic for Special Children, Strasburg, Pennsylvania
  - Greenwood Genetic Center, Greenville, South Carolina
  - University of Utah and Primary Children's Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No